CLINICAL TRIAL: NCT07026370
Title: The China Pulmonary Health Study: Baseline Survey, and Follow-up Investigation
Brief Title: China Pulmonary Health Study
Acronym: CPHS
Status: Active, not recruiting | Type: Observational
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Jieping LEI, Ph.D., Ph.D., China-Japan Friendship Hospital
Other Study IDs: 2022-ZHCH330-01; 2023FY100602 (Other Grant/Funding Number: Ministry of Science and Technology of China); 2016YFC1303900 (Other Grant/Funding Number: Ministry of Science and Technology of China); 201002008 (Other Grant/Funding Number: Ministry of Health of China)
Record Dates: First submitted 2025-05-30; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Chronic Respiratory Diseases; Cardiovascular and Cerebrovascular Diseases; Malignant Tumors; Endocrine and Metabolic Diseases; Multimorbidities
Keywords: Multimorbidities; Epidemiological survey; Cohort; Population medicine
MeSH Terms: conditions — Cerebrovascular Disorders; Neoplasms; Metabolic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The China Pulmonary Health Study (CPHS) was a large-scale epidemiological survey designed to investigate the pulmonary health of Chinese adults aged 20 years or older leveraging a multistage stratified sampling scheme between 2011 and 2014 in mainland China. Briefly, a total number of 57,779 local residents were recruited from 10 representative provinces and municipalities and were invited to participate in the study. A final number of 50,991 adults who met the major inclusion criteria could be considered in further analyses.

In order to investigate the changes of pulmonary health and disease status (e.g. occurrence and development of chronic respiratory diseases and other important relevant multimorbidities, lung function indices, etc.) and corresponding impact factors in the CPHS study population, we plan to initiate the first round of follow-up investigation in 2025 and 2026, i.e. 10-15 years after the baseline survey.

ELIGIBILITY:
Inclusion Criteria:

* (1) the individuals who participated in the CPHS baseline survey;
* (2) their ID number and phone number are available;
* (3) sign the informed consent.

Exclusion Criteria:

* (1) incapable of taking pre- and post-bronchodilator spirometry tests;
* (2) request to withdraw the informed consent;
* (3) terminate due to medical or ethical considerations judged by the investigators and/or ethics committee.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total number of 50,991 adults aged 20 years or older from 10 representative provinces and municipalities of China participated in the CPHS baseline survey between 2011 and 2014. In the follow-up investigation, ideally all the baseline participants should be contacted.
Sampling Method: Non-Probability Sample
Enrollment: 50991 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Occurrence of multimorbidities | Since baseline survey till year 2025 and 2026 (the first round of follow-up investigation of CPHS)
  Occurrence of chronic respiratory diseases, cardiovascular and cerebrovascular diseases, malignant tumors, and/or metabolic diseases, etc.

SECONDARY OUTCOMES:
Changes of lung function, forced expiratory volume in one second (FEV1) | Since baseline survey till year 2025 and 2026 (the first round of follow-up investigation of CPHS)
  Changes of pre- and post-bronchodilator spirometry test indices, FEV1
Changes of lung function, forced vital capacity (FVC) | Since baseline survey till year 2025 and 2026 (the first round of follow-up investigation of CPHS)
  Changes of pre- and post-bronchodilator spirometry test indices, FVC
Changes of lung function, FEV1/FVC | Since baseline survey till year 2025 and 2026 (the first round of follow-up investigation of CPHS)
  Changes of pre- and post-bronchodilator spirometry test indices, FEV1/FVC
Changes of lung function, the percentage of measured FEV1 value to the predicted value (FEV1%pred) | Since baseline survey till year 2025 and 2026 (the first round of follow-up investigation of CPHS)
  Changes of pre- and post-bronchodilator spirometry test indices, FEV1%pred

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang C, Xu J, Yang L, Xu Y, Zhang X, Bai C, Kang J, Ran P, Shen H, Wen F, Huang K, Yao W, Sun T, Shan G, Yang T, Lin Y, Wu S, Zhu J, Wang R, Shi Z, Zhao J, Ye X, Song Y, Wang Q, Zhou Y, Ding L, Yang T, Chen Y, Guo Y, Xiao F, Lu Y, Peng X, Zhang B, Xiao D, Chen CS, Wang Z, Zhang H, Bu X, Zhang X, An L, Zhang S, Cao Z, Zhan Q, Yang Y, Cao B, Dai H, Liang L, He J; China Pulmonary Health Study Group. Prevalence and risk factors of chronic obstructive pulmonary disease in China (the China Pulmonary Health [CPH] study): a national cross-sectional study. Lancet. 2018 Apr 28;391(10131):1706-1717. doi: 10.1016/S0140-6736(18)30841-9. Epub 2018 Apr 9. PMID 29650248
- [Background] Huang K, Yang T, Xu J, Yang L, Zhao J, Zhang X, Bai C, Kang J, Ran P, Shen H, Wen F, Chen Y, Sun T, Shan G, Lin Y, Xu G, Wu S, Wang C, Wang R, Shi Z, Xu Y, Ye X, Song Y, Wang Q, Zhou Y, Li W, Ding L, Wan C, Yao W, Guo Y, Xiao F, Lu Y, Peng X, Zhang B, Xiao D, Wang Z, Chen Z, Bu X, Zhang H, Zhang X, An L, Zhang S, Zhu J, Cao Z, Zhan Q, Yang Y, Liang L, Tong X, Dai H, Cao B, Wu T, Chung KF, He J, Wang C; China Pulmonary Health (CPH) Study Group. Prevalence, risk factors, and management of asthma in China: a national cross-sectional study. Lancet. 2019 Aug 3;394(10196):407-418. doi: 10.1016/S0140-6736(19)31147-X. Epub 2019 Jun 20. PMID 31230828
- [Background] Xiao D, Chen Z, Wu S, Huang K, Xu J, Yang L, Xu Y, Zhang X, Bai C, Kang J, Ran P, Shen H, Wen F, Yao W, Sun T, Shan G, Yang T, Lin Y, Zhu J, Wang R, Shi Z, Zhao J, Ye X, Song Y, Wang Q, Hou G, Zhou Y, Li W, Ding L, Wang H, Chen Y, Guo Y, Xiao F, Lu Y, Peng X, Zhang B, Wang Z, Zhang H, Bu X, Zhang X, An L, Zhang S, Cao Z, Zhan Q, Yang Y, Liang L, Liu Z, Zhang X, Cheng A, Cao B, Dai H, Chung KF, He J, Wang C; China Pulmonary Health Study Group. Prevalence and risk factors of small airway dysfunction, and association with smoking, in China: findings from a national cross-sectional study. Lancet Respir Med. 2020 Nov;8(11):1081-1093. doi: 10.1016/S2213-2600(20)30155-7. Epub 2020 Jun 26. PMID 32598906